CLINICAL TRIAL: NCT05790421
Title: Effect of Foot Muscle Energy Technique in Patients With Diabetic Neuropathy: A Randomized Controlled Trial
Brief Title: Effect of Foot Muscle Energy Technique in Patients With Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Ahmed Magdy Alshimy, Lecturer Of Neurological Physical Therapy - Faculty Of Physical Therapy - October 6 University, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: REC/2111/MTI.PT/2204061
Record Dates: First submitted 2023-03-06; First posted 2023-03-30 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetic neuropathy; Foot muscle energy technique; Isometric muscle strength; Motor nerve conduction velocity study
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants received foot muscle energy techniques and conventional physical therapy program for three sessions/week for 4 weeks, each lasting 30 min
  Interventions: Other: Foot Muscle Energy Technique; Other: Conventional Physical Therapy Program
- Group B (Experimental): Participants received conventional physical therapy program only for three sessions/week for 4 weeks, each lasting 30 min
  Interventions: Other: Conventional Physical Therapy Program

INTERVENTIONS:
Other: Foot Muscle Energy Technique — Starting from the preparation position, at the restriction barrier, the patient is asked to exert a small effort (no more than 20% of available strength) towards plantarflexion, against unyielding resistance, with appropriate breathing. The patient produces isometric effort contracts either gastrocnemius or soleus (depending on whether the knee is unflexed or flexed). This contraction is held for 7-10 seconds together with a held breath. The exercise was repeated until the full range of movement was obtained.
  Other Names: Foot MET
  Arms: Group A
Other: Conventional Physical Therapy Program — Graduated active resisted range of motion exercises for both UL and LL and graduated gait training

SUMMARY:
Foot muscle energy technique and conventional physical therapy program administered in patients with type 2 Diabetic Neuropathy.

DETAILED DESCRIPTION:
Foot muscle energy technique and conventional physical therapy program administered in patients with type 2 Diabetic Neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Participants (males and females) examined with non-insulin-dependent diabetes for ≥10 years determined by neurophysiological measurements were enrolled.
* The participants regularly took their diabetes medications during the assessment and treatment period.
* The use of any sedatives or anticonvulsants was contraindicated for all participants.

Exclusion Criteria:

• Uncontrolled non-insulin dependent diabetes and diagnosed for < 10 years, neural, muscular, and skeletal system deformities; radiculopathy; and psychiatric disorders.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-04-02 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Motor nerve conduction study | 4 weeks
  Assess both tibial and deep peroneal motor nerve conduction velocity.
Toe Strength Dynamometer | 4 weeks
  Assess Isometric muscle strength.

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, El-Sheikh Zayed City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No